CLINICAL TRIAL: NCT05587361
Title: Beta-Adrenergic Modulation of Drug Cue Reactivity: Neural and Behavioral Mechanisms
Brief Title: Beta-Adrenergic Modulation of Drug Cue Reactivity
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oklahoma (Other)
Collaborators: Oklahoma State University Center for Health Sciences (Other); Duke University (Other); National Institute on Drug Abuse (NIDA) (NIH); National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2022005-OSU-CHS; 1R01DA053342-01A1 (NIH)
Record Dates: First submitted 2022-10-03; First posted 2022-10-20 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Tobacco Use Disorder; Nicotine Dependence; Cigarette Smoking
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking | interventions — Propranolol; Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Placebo Patch/Placebo Propranolol (Placebo Comparator): Placebo Nicotine Patch Placebo Propranolol
  Interventions: Drug: Placebo Propranolol; Drug: Placebo Patch
- Placebo Patch/Active Propranolol (Experimental): Placebo Nicotine Patch Active Propranolol (40 mg, immediate release)
  Interventions: Drug: Propranolol; Drug: Placebo Patch
- Active Patch/Placebo Propranolol (Experimental): Active Nicotine Patch (14 mg) Placebo Propranolol
  Interventions: Drug: Nicotine Patch; Drug: Placebo Propranolol
- Active Patch/Active Propranolol (Experimental): Active Nicotine Patch (14 mg) Active Propranolol (40 mg, immediate release)
  Interventions: Drug: Propranolol; Drug: Nicotine Patch

INTERVENTIONS:
Drug: Propranolol — Propranolol Capsule; 40 mg IR
  Arms: Active Patch/Active Propranolol; Placebo Patch/Active Propranolol
Drug: Nicotine Patch — Nicotine Patch; 14 mg
  Arms: Active Patch/Active Propranolol; Active Patch/Placebo Propranolol
Drug: Placebo Propranolol — Placebo Capsule, no active ingredients
  Arms: Active Patch/Placebo Propranolol; Placebo Patch/Placebo Propranolol
Drug: Placebo Patch — Placebo Patch, no active ingredients
  Arms: Placebo Patch/Active Propranolol; Placebo Patch/Placebo Propranolol

SUMMARY:
This study is designed to investigate the effects of a beta-adrenergic antagonist (Propranolol; 40 mg IR) and nicotine patch (14 mg) administered alone and in combination on neurobiological and behavioral responses to smoking cues in ongoing cigarette smokers. This is a basic experimental study in humans and participants will not take these medications for an extended period or make a cessation attempt as part of their involvement in this research project.

DETAILED DESCRIPTION:
Cigarette use remains a serious public health problem in the United States and worldwide. Effective pharmacological interventions for smoking cessation exist, but these medications primarily target nicotine withdrawal and smoking reinforcement. The cues and contexts associated with smoking also play an important role in driving smoking behavior, but evidence is extremely mixed whether existing interventions can effectively attenuate smoking urges and behavior in response to these cues and contexts.

In a previous pilot trial, the investigators demonstrated that propranolol suppressed smoking cue reactivity and brain activation across a constellation of brain regions implicated in nicotine dependence. Here, the investigators seek to extend this work by examining effects when the drug is administered in combination with an established treatment targeting withdrawal and reinforcement (i.e., nicotine patch).

Following consent and screening/baseline activities, participants will attend four neuroimaging appointments each lasting approximately 5 hours. Participants will be fitted with a nicotine or placebo patch, fed a standard meal and then administered propranolol or placebo. Participants will complete questionnaires and have their heart rate/blood pressure monitored throughout the visit. During the MRI scan, participants will be asked to complete both resting scans and task-based scans during which participants will view images of smoking and non-smoking objects and scenes.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy
2. Age 21-60
3. Right-handed using a three-item scale
4. Daily smoker of ≥ 5 cigarettes/day delivering 0.5 mg nicotine (FTC)
5. Smoking regularly for ≥ 1 year, with stable smoking for the past 6 months
6. Afternoon expired Carbon Monoxide (CO) concentration ≥ 6 ppm and/or morning urinary cotinine >100 ng/ml
7. Must identity at least 4 different smoking locations used in a typical week
8. Able to read and understand English

Exclusion Criteria:

1. Inability to attend all required sessions
2. Significant health problems that would preclude active participation
3. Presence of conditions that would make MRI unsafe (e.g. pacemaker) or (e.g. weight and body shape)
4. Current use of psychoactive medications/drugs as indicated by self-report or urine screen
5. Positive breath alcohol concentration
6. Pregnant, breastfeeding, or planning to become pregnant during the course of the study (females)
7. Problems with vision that cannot be corrected with contacts or glasses
8. Current regular use of smokeless tobacco, smoking cessation medications, or other nicotine containing products (e.g. electronic cigarettes)
9. Current use of beta-adrenergic medications (e.g. beta-blockers) or other blood pressure medications
10. Systolic blood pressure < 90 mmHg or diastolic blood pressure < 60 mmHg (sitting or standing)
11. Abnormal EKG
12. Presence of severe anemia
13. Presence of electrolyte imbalance that could impact blood pressure
14. Presence of any other contraindications for propranolol or nicotine patch (e.g. cardiovascular disease, bronchial asthma, prior allergic reactions, diabetes)

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-11-26 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Cue-Provoked Craving Ratings | Approximately 4-5 hours
  Self-reported smoking urges in response to smoking and non-smoking cues during magnetic resonance imaging (MRI) scan. Scores range from 0 to 10 with higher values indicating increased craving for cigarettes.
Blood-Oxygen Level Dependent (BOLD) Activation to Smoking Cues | Approximately 4-5 hours
  Blood-Oxygen Level Dependent (BOLD) Contrast (Smoking-Neutral) in Anterior Hippocampus, Amygdala, Dorsal Anterior Insula, Medial Prefrontal Cortex, Posterior Cingulate Cortex and Ventral Striatum
Association between Smoking Urge and Brain Activation | Approximately 4-5 hours
  Indices of covariation between cue-provoked craving BOLD activation to smoking cues
Hippocampus-Amygdala connectivity to smoking cues | Approximately 4-5 hours
  Index of connectivity between these brain regions
Medial Prefrontal Cortex and Posterior Cingulate Cortex connectivity | Approximately 4-5 hours
  Index of connectivity between these brain regions
Association between Smoking Urge and Brain Connectivity | Approximately 4-5 hours
  Indices of covariation between cue-provoked craving BOLD activation to smoking cues

CONTACTS AND LOCATIONS:
Overall Officials: Jason A Oliver, PhD, Principal Investigator — University of Oklahoma
Locations (1):
- Hardesty Center for Clinical Research and Neuroscience, Tulsa, Oklahoma, United States